CLINICAL TRIAL: NCT05076929
Title: Assessment of Ultrasonographic Measurement of Inferior Vena Cava Collapsibility Index in Prediction of Hypotension Associated With Tourniquet Release in Total Knee Replacement Surgeries Under Spinal Anesthesia
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mona Ammar, Assistant Professor, Ain Shams University
Other Study IDs: MS 292/ 2021
Record Dates: First submitted 2021-09-26; First posted 2021-10-13 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Fluid Hypovolemia, Cerebrospinal
MeSH Terms: conditions — Intracranial Hypotension | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ultrasound — Ultrasonographic measurement of Inferior Vena Cava Collapsibility Index

SUMMARY:
Administration of intravascular fluids is one of the methods to prevent SA-induced hypotension, but empirical intraoperative volume repletion carries the risk of fluid overload during elective surgery. Over fluid resuscitation is associated with organ dysfunction and higher mortality rate , thus, to avoid ineffective or even harmful intravascular volume expansion, it is important to have tools to predict hypotension and fluid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* ASA grade I, II, III
* Age 18 -65 yrs
* Spinal Anesthesia

Exclusion Criteria:

* Patient refusal
* Patient having contraindication of Spinal Anesthesia (infection at the site of injection, spine deformity, coagulation disorders ) .
* Known cardiac, renal, neurological, metabolic, endocrine, psychiatric, respiratory disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total Knee Replacement Surgeries under Spinal Anesthesia
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
mean arterial blood pressure | 15 minutes after tourniquet release

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No